CLINICAL TRIAL: NCT02970240
Title: Cardiopulmonary Exercise Testing as a Diagnostic Tool and a Quantitative Measure of Post-exertional Malaise in Myalgic Encephalopathy/Chronic Fatigue Syndrome
Brief Title: Cardiopulmonary Testing in ME/CFS to Improve Diagnostic Accuracy
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: The Glittre Clinic (Unknown); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Per Ole Iversen, MD, Professor, University of Oslo
Other Study IDs: 2012/571
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome
Keywords: cardiopulmonary exercise testing; inflammation; oxidative status
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Inflammation | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ME/CFS group: Patients with a verified diagnosis of ME/CFS according to the Canada criteria
  Interventions: Procedure: Cardiopulmonary testing
- Fatigue group: Patients with fatigue, but not ME/CFS
  Interventions: Procedure: Cardiopulmonary testing
- Control group: Healthy control persons
  Interventions: Procedure: Cardiopulmonary testing

INTERVENTIONS:
Procedure: Cardiopulmonary testing — A 2-day consecutive testing on an ergometer cycle

SUMMARY:
Circumstantial evidence suggests that patients diagnosed with myalgic encephalopathy/chronic fatigue syndrome (ME/CFS) perform worse on day 2 in a 2-day consecutive cardiopulmonary exercise test (CPET). The aim of this study is to examine if CPET can distinguish between ME/CFS patients and healthy controls.

DETAILED DESCRIPTION:
Myalgic encephalopathy/chronic fatigue syndrome (ME/CFS) leads to a substantial reduction in activity level. Cardiopulmonary exercise testing (CPET) quantifies physical performance, or functional capacity, by direct measurements of the maximal oxygen uptake (VO2max). Functional capacity is the ability of an individual to perform aerobic work as defined by the VO2max, and the assessment of functional capacity reflects the ability to perform activities of daily living that require sustained aerobic metabolism.

To the best of knowledge few robustly designed studies on repeated CPET in ME/CFS are published, and they demonstrated a significant reduction in functional capacity expressed as VO2max and anaerobic threshold. This marked functional decline on the second test has apparently not been described for any other chronic, disabling conditions, and might represent a possible diagnostic tool for ME/CFS; hence the investigators will examine this. In addition they will examine other biological markers (e.g. cytokines and anti-oxidative compounds) before and after the exercise tests to test if the groups can be further distinguished.

The main aim of this study is to evaluate the use of repeated CPET as an objective diagnostic marker of ME/CFS. Specifically the investigators want to address the following questions:

I. Will patients with ME/CFS demonstrate a significant reduction in VO2max compared to healthy individuals? If such a difference can be demonstrated, is it unique for patients with ME/CFS classified according to the strictest criteria compared to others with longstanding fatigue?

II. What is the blood lactate profile before, during and after CPET?

III. Are there any correlations between the decline in VO2max and other biological variables such as markers of oxidative stress, immune dysregulation or metabolic dysfunction?

IV. Is cardiac function impaired among ME/CFS patients as assessed by ecco-cardiography?

Three groups will be included: (i) ME/CFS patients; (ii) patients with fatigue, but not MF/CFS; and (iii) healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ME/CFS according to the Canadian and Fukuda criteria; miid to moderately affected)
* Provide written consent
* Able to perform the test

Exclusion Criteria:

* Not provided written consent
* Unable to perform the test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with ME/CFS
  2. Patients with fatigue but not ME/CFS
  3. Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | At 48 hour
  Measurement of oxygen uptake during ergometer cycling

SECONDARY OUTCOMES:
Lactate accumulation | At 48 hour
  Regular sampling of blood for measurements of lactate
Cytokine profile | At 48 hour
  Regular sampling of blood for measurements of cytokines
Immunophenotyping | At 48 hour
  Regular sampling of blood for measurements of cell surface markers
Cardiac status | At 48 hour
  Measurements of Cardiac function using ecco-cardiography

CONTACTS AND LOCATIONS:
Overall Officials: Per O Iversen, MD, Principal Investigator — University of Oslo
Locations (1):
- Glittre Clinic, Hakadal, Norway

IPD SHARING:
Plan to Share IPD: No